CLINICAL TRIAL: NCT02448758
Title: Cohort of Non-small Cell Lung Cancer With Mutation of the Nord Pas de Calais
Brief Title: Cohort of Non-small Cell Lung Cancer With Mutation of the Nord Pas de Calais (CB(NPC)²)
Acronym: CB(NPC)²
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Oscar Lambret (Other)
Collaborators: University Hospital, Lille (Other); Centre de Biologie Pathologie : Plateforme de Biologie Moléculaire de Lille (Unknown)
Responsible Party: Sponsor
Other Study IDs: CB(NPC)²-1209
Record Dates: First submitted 2014-03-06; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to create a database at the regional level, the principle is to include all patients in whom a mutation was detected from a single platform (Lille). The creation of this regional cohort, smaller than the national cohort of Biomarkers France, will perform a more comprehensive collection of clinical data, and molecular monitoring data of patients included. To increase the completeness of the collection of information, it will not be based on voluntary prescribing clinician but will be largely carried out by CRA dedicated to this activity.

DETAILED DESCRIPTION:
This is a prospective and retrospective study of a population of patients with mutated non-small cell lung cancer in the Nord Pas de Calais. Retrospective cohort will involve patients with main molecular abnormalities, identifiable from molecular biology platform CRRC, except EGFR and KRAS treated from September 2011 to February 2013.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Patient with non-small cell lung cancer
* Detected in the Nord Pas de Calais
* Monitored in the Nord Pas de Calais
* Patient must have signed a non-opposition form to the use of medical data

Exclusion Criteria:

- No identified mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer with mutation of the Nord Pas de Calais
Sampling Method: Non-Probability Sample
Enrollment: 785 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between clinical factors and mutation status | at baseline
  The clinical factors are age, smoking status, occupational and environmental exposure, personal and family background, TNM stage, performance status

SECONDARY OUTCOMES:
Progression-free survival | 3 years
Overall survival | 3 years
Number of patients included in a clinical trial dedicated to a certain type of non-small cell lung cancer with mutation | 3 years
Number of cases per mutation type | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexis CORTOT, MD, PhD, Study Director — CHRU of Lille; Eric Dansin, MD, Study Director — Centre Oscar Lambret
Locations (2):
- France (2):
  - Centre Oscar Lambret, Lille
  - CHRU, Lille